CLINICAL TRIAL: NCT04381962
Title: A Multi-centre Open-label Two-arm Randomised Superiority Clinical Trial of Azithromycin Versus Usual Care In Ambulatory COVID-19 (ATOMIC2)
Brief Title: A Multicentre Open-label Two-arm Randomised Superiority Clinical Trial of Azithromycin Versus Usual Care In Ambulatory COVID19 (ATOMIC2)
Acronym: ATOMIC2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATOMIC2; 2020-001740-26 (EudraCT Number); 282892 (Other: IRAS); 20/HRA/2105 (Other: London-Brent Research Ethics Committee)
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2020-05

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Coronavirus; COVID-19; Azithromycin; Respiratory failure; Mortality; Trial
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Respiratory Insufficiency | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Open label, Two-arm, Randomised Superiority Trial
Masking Description: This is an open-label study. However, while the study is in progress, access to tabular results by allocated treatment allocation will not be available to the research team, patients, or members of the Steering Committee (unless the DSMC advises otherwise).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin (Experimental): Azithromycin 2x250mg capsules to be taken orally once daily for 14 days. The first dose will be within 4 hours of randomisation. This is in addition to standard care as per local hospital advice for those patients with suspected COVID who are not admitted: i.e. symptomatic relief with rest, as-required paracetamol (where appropriate) and advice to seek further medical attention if significant worsening of breathlessness.
  Interventions: Drug: Azithromycin Capsule
- Usual standard care (No Intervention): Standard care as per local hospital advice for those patients with suspected COVID who are not admitted: i.e. symptomatic relief with rest, as-required paracetamol (where appropriate) and advice to seek further medical attention if significant worsening of breathlessness.

INTERVENTIONS:
Drug: Azithromycin Capsule — Azithromycin 500 mg OD PO 14 days
  Arms: Azithromycin

SUMMARY:
A multi-centre open-label two-arm randomised superiority clinical trial of two weeks of oral Azithromycin 500mg once daily versus usual care in adult patients presenting to secondary care with clinically-diagnosed COVID-19 but assessed as appropriate for initial ambulant (outpatient) management, in preventing progression to respiratory failure or death.

DETAILED DESCRIPTION:
Hypothesis: Use of Azithromycin 500 mg once daily for 14 days is effective in preventing and/or reducing the severity of lower respiratory illness of COVID-19 disease at 28 days.

Study design: Multi centre, prospective open label two-arm randomised superiority clinical trial of standard care and Azithromycin with standard care alone for those presenting to hospital with COVID-19 symptoms who are not admitted at initial presentation.

Study setting: Patients being assessed by secondary care NHS hospitals in the UK.

Participants: Adults, ≥18 years of age assessed in an acute hospital with clinical diagnosis of COVID-19 infection and where medically it is decided not to admit the patient and for the patient to be managed on an ambulatory (outpatient) care pathway at their usual residence (home or care home).

Study schedule: Enrolment on day 0. Telephone follow up at day 14 day, and day 28. If admitted between randomisation and day 28, data will be collected until hospital discharge.

Intervention: Azithromycin 500 mg orally once daily for 14 days. The first dose will be within 4 hours of randomisation. This is in addition to standard care as per local hospital advice for those patients with suspected COVID who are not admitted: i.e. symptomatic relief with rest, as-required paracetamol (where appropriate) and advice to seek further medical attention if significant worsening of breathlessness.

Comparator: Standard care as per local hospital advice for those patients with suspected COVID who are not admitted: i.e. symptomatic relief with rest, as-required paracetamol (where appropriate) and advice to seek further medical attention if significant worsening of breathlessness.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged at least 18 years
* Assessed by the attending clinical team as appropriate for initial ambulatory (outpatient) management
* A clinical diagnosis of highly-probable COVID-19 infection (diagnosis by the attending clinical team)
* No medical history that might, in the opinion of the attending clinician, put the patient at significant risk if he/she were to participate in the trial
* Able to understand written English (for the information and consent process) and be able to give informed consent

Exclusion Criteria:

* Known hypersensitivity to any Macrolide including Azithromycin, Ketolide antibiotic, or the excipients including an allergy to soya or peanuts.
* Known fructose intolerance, glucose-galactose malabsorption or sucrose-isomaltase-insufficiency
* Currently on a Macrolide antibiotic (Clarithromycin, Azithromycin, Erythromycin, Telithromycin, Spiramycin)
* On any SSRI (Selective Serotonin Reuptake Inhibitor)
* Elevated cardiac troponin at initial assessment suggestive of significant myocarditis (if clinically the clinical team have felt it appropriate to check the patient's troponin levels)
* Evidence of QTc prolongation: QTc>480ms
* Significant electrolyte disturbance (e.g. hypokalaemia K+<3.5 mmol/L)
* Clinically relevant bradycardia (P<50 bpm), non-sustained ventricular tachycardia or unstable severe cardiac insufficiency
* Currently on hydroxychloroquine or chloroquine

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Proportion progressing to respiratory failure or death (all clinically-diagnosed participants) | Determined at day 28 from randomisation.
  Efficacy will be determined through differences in the proportion with either death or admission with respiratory failure requiring level 2 ventilation (NIV/CPAP/nasal high-flow) or level 3 (invasive mechanical ventilation) in the 28 days from randomisation.

SECONDARY OUTCOMES:
Proportion progressing to respiratory failure or death (SARS-CoV-2 PCR positive) | Determined at day 28 from randomisation.
  Efficacy will be determined through differences in the proportion with either death or admission with respiratory failure requiring level 2 ventilatory support (NIV/CPAP/nasal high-flow) or level 3 (invasive mechanical ventilation) in the 28 days from randomisation using a retrospective analysis of COVID-19 oropharyngeal swabs for those who had one taken at time of randomisation.
All cause mortality | Ascertain data at 28 days after randomisation.
  Data on vital status (alive / dead, with date and presumed cause of death if appropriate)
Proportion progressing to pneumonia. | Ascertain this information at time of pneumonia diagnosis, or at 28 days after randomisation (whichever is sooner)
  Progression to pneumonia as diagnosed by chest x-ray (or CT thorax), with compatible clinical findings, if no pneumonia is present at time of enrolment. To be diagnosed by a medically qualified doctor and data obtained from review of case-notes and relevant radiology.
Proportion progressing to severe pneumonia | Ascertain this information at time of pneumonia diagnosis, or at 28 days after randomisation (whichever is sooner)
  Evolution of pneumonia, as diagnosed by chest x-ray or CT thorax, if pneumonia is present at time of enrolment. To be diagnosed by a medically qualified doctor and data obtained from review of case-notes and relevant radiology. Severe pneumonia is defined as BTS CURB-65 score of 3-5.
Peak severity of illness | Ascertain from day 14 and day 28 telephone call and from retrospective ePR/medical notes data at 28 days after randomisation.
  The 9-point ordinal scoring system is described in the protocol reflects the severity of respiratory illness. The maximum severity score during the entire study period will be compared.
Safety and tolerability | Emergent data collection days 0-28 and elicit proactively at day 14 and day 28 post randomisation.
  Serious adverse events and concomitant medications. Record at enrolment, emergently during study period and proactively elicit at day 14 and at day 28.

OTHER OUTCOMES:
Mechanistic analysis of blood and nasal biomarkers if available | Samples to be collected prospectively at baseline and again if patient admitted, to be taken as soon as possible and within 72 hours of admission if possible.
  The following samples may be taken. Blood for serum, Tempus tube (whole blood RNA), EDTA tubes (PBMC), nasal brush to be placed immediately into RNA lysis buffer (for subsequent PCR and transcriptomic analysis). Includes assessment of mycoplasma prevalence for subgroup analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Little, MD PhD, Study Chair — University of Southampton
Locations (5):
- United Kingdom (5):
  - Horton General Hospital, Banbury, Oxfordshire
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - Ninewells Hospital, Dundee, Scotland
  - Birmingham City Hospital, Birmingham
  - Sandwell General Hospital, West Bromwich

REFERENCES:
- [Background] Hinks TSC, Barber VS, Black J, Dutton SJ, Jabeen M, Melhorn J, Rahman NM, Richards D, Lasserson D, Pavord ID, Bafadhel M. A multi-centre open-label two-arm randomised superiority clinical trial of azithromycin versus usual care in ambulatory COVID-19: study protocol for the ATOMIC2 trial. Trials. 2020 Aug 17;21(1):718. doi: 10.1186/s13063-020-04593-8. PMID 32807209
- [Derived] Hinks TSC, Cureton L, Knight R, Wang A, Cane JL, Barber VS, Black J, Dutton SJ, Melhorn J, Jabeen M, Moss P, Garlapati R, Baron T, Johnson G, Cantle F, Clarke D, Elkhodair S, Underwood J, Lasserson D, Pavord ID, Morgan S, Richards D. Azithromycin versus standard care in patients with mild-to-moderate COVID-19 (ATOMIC2): an open-label, randomised trial. Lancet Respir Med. 2021 Oct;9(10):1130-1140. doi: 10.1016/S2213-2600(21)00263-0. Epub 2021 Jul 9. PMID 34252378
- See also: ATOMIC2 homepage — https://atomic2.octru.ox.ac.uk